CLINICAL TRIAL: NCT02997462
Title: Monocyte Phenotypic Changes in Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Scott L. Hummel, Associate Professor, University of Michigan
Other Study IDs: HUM00049322
Record Dates: First submitted 2012-03-19; First posted 2016-12-20 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Decompensated Heart Failure
Keywords: Monocyte; Oxidative Stress; Endothelial Function; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for cytokine measures
  Blood samples for monocyte cell surface marker and functional phenotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure: Heart Failure patients admitted to the ICU or Heart Failure Service.
  No changes in service-directed plan of care for patients.
- Healthy Control: Healthy, age-matched controls.

SUMMARY:
There are many treatments that can improve how long and how well people live with heart failure when they are outside the hospital. However, the investigators know less about how to effectively treat hospitalized heart failure patients so that they do not have to return to the hospital after they go home. Part of the problem is that the investigators don't understand all of the causes of worsening heart failure.

Previous studies by other researchers suggest that white blood cells called monocytes are over-active in heart failure. Under normal conditions monocytes help fight infections in the body, but over-active monocytes release chemicals that could cause abnormal function of the heart and blood vessels. The investigators' research group believes that over-active monocytes may be an important reason that heart failure worsens before hospitalization.

In this study the investigators will collect blood samples on the day a patient comes into the hospital, the day they return home, and the day they come back to the clinic for a follow-up appointment. The investigators will measure the inflammation in the bloodstream and the activity of monocytes from the patients' blood to see if there are changes in these measurements as heart failure improves. The investigators will also call each patient several times after they return home to ask questions about how they are doing.

DETAILED DESCRIPTION:
With over 5 million Americans having heart failure (HF) today and an incidence approaching 10 per 1000 population among persons over the age of 65, HF is a major source or morbidity and mortality and a significant public health concern facing developed nations. In the US, decompensated heart failure is the most common reason for hospital admission among persons older than 65. Yet despite significant advances in the treatment of chronic heart failure, currently there are very few evidence-based strategies to treat acutely decompensated heart failure. The incidence of heart failure will likely continue to rise with the increasing prevalence of HF risk factors (advanced age, hypertension, obesity, diabetes, and other metabolic diseases). Accordingly, substantial efforts are underway to identify and treat populations at risk and to understand the molecular drivers of this heterogeneous disease.

The investigators understanding of the pathophysiology of heart failure has evolved from a 'cardiocentric' view focused on mechanical dysfunction to a more global view. Heart failure is now understood as a complex blend of structural, functional, and neurohormonal abnormalities manifested both locally and systemically. More recently, several groups have demonstrated abnormalities in the inflammatory cascade associated with both the initiation and the progression of heart failure. The innate immune system appears to modulate the inflammatory component of HF through several mechanisms including the production of inflammatory cytokines (tumor necrosis factor-α,TNFα; interleukin-6, IL6), reactive oxygen species, activation of the complement system, as well as through functional modification of endothelial cells and myeloid cell trafficking.

Monocytes and macrophages are two of the key myeloid mediators of acute and chronic inflammatory responses. Myeloid dysregulation has been implicated in the pathogenesis of diverse diseases including diabetes, tumor metastasis, pulmonary fibrosis, myocardial infarction, and atherosclerosis. Accumulating evidence suggests that myeloid subsets have distinct functional properties reflecting their polarization patterns and their interaction with the local microenvironment. As a framework to study their role in models of clinical diseases, myeloid populations have been broadly categorized as "inflammatory" and "anti-inflammatory" based on specific surface markers, cytokine potential, and other functional properties.

Although the role of myeloid populations in inflammatory disease is now appreciated, the molecular mechanisms linking these cells to clinical heart failure syndromes remain largely unknown. The investigators hypothesize that distinct myeloid subsets drive different phases of acute and chronic heart failure syndromes, and that identification of these subsets and their functional properties will provide further insight into the pathophysiology of clinical heart failure.

In order to initially characterize the roles that monocytes play across the spectrum of heart failure, the investigators will obtain whole-blood samples from acutely decompensated patients on the date of hospitalization, the date of transfer from the intensive care unit (ICU) to the general-care telemetry floor (if relevant), the date of hospital discharge, and at their first outpatient follow-up visit. Subjects will be recruited from the University of Michigan inpatient heart failure service, which admits approximately 75 patients for decompensated heart failure each month. Once the samples are obtained, the investigators will perform flow cytometry to characterize monocyte subsets and their flux in response to treatment. The investigators will also look at the production of reactive oxygen species by monocytes and will examine how cytokines and chemokines skew monocyte population subsets and their gene expression profiles. The investigators will also investigate the energetic state and flux (aerobic vs. anaerobic metabolic status) of the monocytes.

ELIGIBILITY:
Inclusion Criteria: Heart Failure Patients:

* 18 years of age or older
* Patients must be diagnosed with heart failure
* Patients must be hospitalized at the University of Michigan Hospital for treatment of heart failure symptoms.

Exclusion Criteria: Heart Failure Patients:

* Heart attack or other active problem with coronary artery disease
* Severe kidney failure or need for dialysis
* An active infection or inflammatory condition
* A need for treatment that affects the immune system (e.g. systemic steroids, immunomodulatory therapies)
* A planned surgery during this hospital admission, including heart transplant or other heart surgery

Inclusion Criteria: Healthy Control Patients:

- Must be greater than or equal to 65 years of age

Exclusion Criteria: Healthy Control Patients:

* Diabetes
* High blood pressure
* Active cancer
* Heart disease
* Lung disease
* Liver disease
* Kidney disease
* Active smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure inpatients and age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change in IL-6 between hospital admission and discharge | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Cytokine

SECONDARY OUTCOMES:
Lys6c Hi and Lo, Mannose Receptor | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Cell Surface Markers
IL-10, IL-13 | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Cytokine
Gene Expression (iNOS, CCL2, Ym1, Fizz, VEGF, MMP2/9) | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Monocyte gene expression
microRNA | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  miR155, let7, mir-33a
Monocyte/macrophage morphology | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Macrophages/monocytes will be classified based on their morphology
Serum F-2 Isoprostanes | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Oxidative stress marker
TNF-alpha | All scheduled blood draws - hospital admission, discharge (3-14 days after admission), and first post-discharge appointment (5-10 days following discharge)
  Marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hummel, MD MS, Principal Investigator — University of Michigan; Adam Stein, MD, Principal Investigator — University of Michigan; Sascha Goonewardena, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Seidler S, Zimmermann HW, Bartneck M, Trautwein C, Tacke F. Age-dependent alterations of monocyte subsets and monocyte-related chemokine pathways in healthy adults. BMC Immunol. 2010 Jun 21;11:30. doi: 10.1186/1471-2172-11-30. PMID 20565954
- [Background] Polidori MC, Pratico D, Savino K, Rokach J, Stahl W, Mecocci P. Increased F2 isoprostane plasma levels in patients with congestive heart failure are correlated with antioxidant status and disease severity. J Card Fail. 2004 Aug;10(4):334-8. doi: 10.1016/j.cardfail.2003.11.004. PMID 15309701
- [Background] Colombo PC, Banchs JE, Celaj S, Talreja A, Lachmann J, Malla S, DuBois NB, Ashton AW, Latif F, Jorde UP, Ware JA, LeJemtel TH. Endothelial cell activation in patients with decompensated heart failure. Circulation. 2005 Jan 4;111(1):58-62. doi: 10.1161/01.CIR.0000151611.89232.3B. Epub 2004 Dec 20. PMID 15611373
- [Background] Levine B, Kalman J, Mayer L, Fillit HM, Packer M. Elevated circulating levels of tumor necrosis factor in severe chronic heart failure. N Engl J Med. 1990 Jul 26;323(4):236-41. doi: 10.1056/NEJM199007263230405. PMID 2195340
- [Background] Deswal A, Petersen NJ, Feldman AM, Young JB, White BG, Mann DL. Cytokines and cytokine receptors in advanced heart failure: an analysis of the cytokine database from the Vesnarinone trial (VEST). Circulation. 2001 Apr 24;103(16):2055-9. doi: 10.1161/01.cir.103.16.2055. PMID 11319194
- [Background] Mann DL, McMurray JJ, Packer M, Swedberg K, Borer JS, Colucci WS, Djian J, Drexler H, Feldman A, Kober L, Krum H, Liu P, Nieminen M, Tavazzi L, van Veldhuisen DJ, Waldenstrom A, Warren M, Westheim A, Zannad F, Fleming T. Targeted anticytokine therapy in patients with chronic heart failure: results of the Randomized Etanercept Worldwide Evaluation (RENEWAL). Circulation. 2004 Apr 6;109(13):1594-602. doi: 10.1161/01.CIR.0000124490.27666.B2. Epub 2004 Mar 15. PMID 15023878
- [Background] Aukrust P, Ueland T, Lien E, Bendtzen K, Muller F, Andreassen AK, Nordoy I, Aass H, Espevik T, Simonsen S, Froland SS, Gullestad L. Cytokine network in congestive heart failure secondary to ischemic or idiopathic dilated cardiomyopathy. Am J Cardiol. 1999 Feb 1;83(3):376-82. doi: 10.1016/s0002-9149(98)00872-8. PMID 10072227